CLINICAL TRIAL: NCT02895490
Title: Using Communication Training to Promote Employment Retention Among Cancer Survivors
Brief Title: Communication Training in Promoting Employment Retention Among Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant ended/funding unavailable
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-14021; NCI-2013-02478 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HM14021 (Other: IRB No.); MCC-14021 (Other: Virginia Commonwealth University/Massey Cancer Center)
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (DVD) (Experimental): Patients receive a DVD containing educational information about patients' legal rights in the workplace and communication skills demonstrated through four scenarios depicting a variety of employer-employee communication challenges for patients, provided by LINC group.
  Interventions: Other: educational intervention; Other: communication skills training; Other: questionnaire administration; Other: quality-of-life assessment
- Arm II (control) (Active Comparator): Patients receive information about the LINC group.
  Interventions: Other: educational intervention; Other: questionnaire administration; Other: quality-of-life assessment

INTERVENTIONS:
Other: educational intervention — Receive a DVD containing educational information and communication skills
  Other Names: intervention, educational
  Arms: Arm I (DVD)
Other: communication skills training — Receive a DVD containing educational information and communication skills
  Arms: Arm I (DVD)
Other: educational intervention — Receive information about the LINC group
  Other Names: intervention, educational
  Arms: Arm II (control)
Other: questionnaire administration — Ancillary studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This randomized clinical trial studies communication training in promoting employment retention among cancer patients. Communication training may improve patient-employer communication and increase the likelihood that cancer patients will remain employed, reduce patients' time away from work, and increase workplace accommodations that enable patients to balance treatment and work.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate the efficacy of the DVD intervention to a) increase patients' knowledge of their legal rights in the workplace, b) improve patient perceptions of workplace communication about the impact of cancer treatment and ongoing surveillance, and c) increase the number of requested and received workplace accommodations.

II. Compare employment status (employed vs non-employed) between the treatment and control arms.

III. Compare weekly hours of work between the treatment and control arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

Arm I: Patients receive a DVD containing educational information about patients' legal rights in the workplace and communication skills demonstrated through four scenarios depicting a variety of employer-employee communication challenges for patients, provided by the Legal Information Network for Cancer (LINC) group.

Arm II: Patients receive information about the LINC group

After completion of study, patients are followed up at 4, 12, and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new, primary diagnosis of a solid tumor
* Employed full- or part-time at the time of enrollment
* English-speaking
* Able to participate in telephone interviews
* Able to view a 1-hour DVD
* Patients must have a treatment plan that includes chemotherapy and be within 2 weeks of initiating chemotherapy

Exclusion Criteria:

* Patients with prior cancer except non-melanoma skin cancer

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Changes in perceived self-efficacy pre-intervention and post-intervention. | Baseline to up to 52 weeks
  Modify the Perceived Efficacy in Patient-Physician Interactions (PEPPI) to measure patient confidence in talking with their employer. The revised version will focus on patients' level of confidence in discussing employer accommodation and seeking support from their employer. The PEPPI is a brief ten-item measure that asks patients to rate on a Likert scale their confidence in communicating. It is a widely used measure with strong psychometric properties anchored at 5 - "very confident" and 1 - "not at all confident." Thus, the investigators plan to evaluate communication self-efficacy before and after patients in the experimental group view the DVD to explore changes in perceived self-efficacy as a result of communication training. The investigators will compare this change with changes in the control group patients' perceived self-efficacy by matching the timing of the pre-post administration of the measure in both groups.
Compare requested pre-intervention measures to received post-intervention measures. | Baseline to up to 52 weeks
  During the baseline (pre-intervention) interview patients will answer these questions about specific workplace topics the patients is interested in discussing with their employer, such as available accommodations. During the interviews, each patient will complete a matched questionnaire asking about whether or not they discussed these topics. A score of "1" on the pre-intervention measure indicates patients wanted to discuss the item and the same score on the post-interventions measures indicates that this topic was discussed. A score of "0" in the post-intervention measure indicates that this expectation was not met.
Compare longitudinal changes in knowledge scale before and after combination information and communication skills training. | Baseline to up to 52 weeks
  To aid knowledge acquisition, the investigators have linked didactic teaching with video recorded scenarios exemplifying use of knowledge and skills to achieve increased knowledge. The investigators have developed a knowledge measure and in collaboration with Dr. Dumenci will rigorously test the scale. The investigators will then use this scale to determine whether patients' knowledge improves as a result of the combination of information and communication skills training proposed in this intervention. Therefore, knowledge will be measured before the intervention and after the intervention. The investigators will then compare the experimental and control groups' longitudinal changes in knowledge.

SECONDARY OUTCOMES:
Compare the amount of weekly hours worked between treatment and control arms. | Baseline to up to 52 weeks
  Compare weekly hours of work between the treatment and control arms
Compare the amount of employed vs non-employed subjects between treatment and control arms. | Baseline to up to 52 weeks
  Compare employment status (employed vs non-employed) between the treatment and control arms.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brown, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States